CLINICAL TRIAL: NCT04255706
Title: Evaluation of Repeatability in Measurements of Two Swept-source Optical Coherence Tomography (Ss-OCT) Biometers and One Optical Low Coherence Reflectometry (OLCR) Biometer
Brief Title: Repeatability in Measurements of Two ssOCT and One OLCR Biometer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of the Ophthalmology Department, and Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANT
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Cataract Senile
Keywords: ss-OCT; OLCR; biometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Biometric measurement repeatability (Other): Biometric measurements will be performed in all patients
  Interventions: Device: biometric measurement IOLMaster 700; Device: biometric measurement Lenstar LS 700; Device: biometric measurement Anterion Heildelberg

INTERVENTIONS:
Device: biometric measurement IOLMaster 700 — Three biometric measurements will be performed with 3 devices for all the patients included
Device: biometric measurement Lenstar LS 700 — Three biometric measurements will be performed with 3 devices for all the patients included
Device: biometric measurement Anterion Heildelberg — Three biometric measurements will be performed with 3 devices for all the patients included

SUMMARY:
Achieving high accuracy and precision in ocular biometry has become primordial for cataract surgery, due to the shift of cataract surgery from a rehabilitation procedure to a refractive one.

Aim of this study is to determine the repeatability of ocular biometric parameters obtained using three biometry devices, two ss-OCT biometers and an OLCR device.

DETAILED DESCRIPTION:
Accurate and repeatable biometric measurements are essential in providing an optimal refractive outcome.

ss-OCT biometry uses a tunable wavelength laser source to scan the eye, this technology showing its superiority through better signal-to-noise ratio, the wavelength light source being projected into the eye, one at a time; thus improving tissue penetration.

This a prospective observational study that would include patients which attended pre-surgical examination. A written informed consent will be obtained from each patient.

Only one eye from each patient will be included in the study. All patients included in the study will undergo biometric measurements in a random fashion with the three devices (IOLMaster 700, Lenstar LS 700 and Anterion Heildelberg). Each patient will be measured three times with each device and between the measurements they will be asked to blink or keep their eyes closed for tear film recovery and to avoid fatigue. Scans that pass the quality requirement of each device will be taken for analysis.

ELIGIBILITY:
Inclusion Criteria:

* 40 years old or above
* age-related cataract

Exclusion Criteria:

* patients with dense cataract or corneal pathology that would significantly influence biometric measurements
* nystagmus or pathologies that would affect patient fixation
* pregnancy- for women in reproductive age a pregnancy test will be performed.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of repeatability between two ss-OCT and one OLCR biometry device | 8 months
  Repeatability coefficient (within subject standard deviation - SD) and coefficient of variation between two ss-OCT and the OLCR biometry device will be calculated for all the parameters (axial length, keratometry, anterior chamber depth, lens thickness)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof, Principal Investigator — VIROS, Hanusch Hospital Vienna
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fisus AD, Hirnschall ND, Ruiss M, Pilwachs C, Georgiev S, Findl O. Repeatability of 2 swept-source OCT biometers and 1 optical low-coherence reflectometry biometer. J Cataract Refract Surg. 2021 Oct 1;47(10):1302-1307. doi: 10.1097/j.jcrs.0000000000000633. PMID 33770018